A clinical prospective study to validate a risk scoring model integrated preoperative immune-inflammatory indicators, tumor markers and imaging examination for the lymph node metastasis of

gastric cancer before surgery (DJY004 Trail)

**Edition Number: 1.0** 

**Edition Generation Date:** Jul 1, 2023

**Principal Investigator: Jingyu Deng** 

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## **Statistical Analysis Plan**

Continuous variables will be reported as either mean ± standard deviation or median (interquartile range). Categorical variables will be analyzed using the Chi-square test or Fisher's exact test, while continuous variables will be assessed using the T test or Mann–Whitney U test. The model's sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) will be calculated, along with evaluating the consistency between actual occurrences of postoperative hepatic metastases and the model's predicted results. To assess the calibration ability of the risk scoring model, the area under the receiver operating characteristic curve (AUROC) will be computed. Statistical significance will be set at a p-value threshold of 0.05. All statistical analyses will be conducted using SPSS 26.0 software and R software.